CLINICAL TRIAL: NCT04696562
Title: The Effect of Deep Breathing Exercise Applied With Triflo on Dyspnea, Anxiety and Quality of Life in Patients Treated for COVID-19: Randomized Controlled StudyPatients Treated for COVID-19: A Randomized Controlled Study
Brief Title: The Effect of Deep Breathing Exercise on Dyspnea, Anxiety and Quality of Life in Patients Treated for COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hatice ÖNER CENGİZ, Lecturer PhD., Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OCengiz
Record Dates: First submitted 2020-12-30; First posted 2021-01-06 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: COVID-19; Breathing Exercises; Dyspnea; Anxiety; Quality of Life
MeSH Terms: conditions — COVID-19; Dyspnea; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This single-centered, randomized controlled study will be held in Ankara city hospital in Turkey. The investigators used the G*Power (Version 3.1.9) test to determine the sample size. Participants included patients who treated in hospital for covid-19 who fulfilled the inclusion criteria and agreed to participate.
  Randomized block assignment was used to assign 44 patients to the intervention group (n = 22) and the control group (n = 22). The investigators did block randomization, via a computer program (sealed envelope, https://www.sealedenvelope.com/ , randomization code: 34780089372265).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group is the group in which the investigors applied deep breathing exercises with triflo.
  Interventions: Behavioral: Deep Breathing Exercise with Triflo
- Control group (No Intervention): The control group is the group that receives standard clinical care.

INTERVENTIONS:
Behavioral: Deep Breathing Exercise with Triflo — The investigators will do deep breathing exercises 5-10 times an hour with the triflo device.
  Arms: Intervention group

SUMMARY:
The world is facing an extremely important global epidemic. Coronavirus disease 2019 (COVID-19) epidemic, which first appeared in Wuhan, China in late 2019 and rapidly affected all countries of the world, was declared as a pandemic by the World Health Organization (WHO) on March 11, 2020. Coronavirus disease 2019 affects both the upper (i.e. sinuses, nose and throat) and lower (i.e. trachea and lungs) airways, causes respiratory tract diseases ranging from asymptomatic or cold to more severe lung diseases (Acute Respiratory Distress Syndrome-ARDS). COVID-19 has many symptoms (i.e. fever, loss of appetite). In cases where the disease has a more severe course, in addition to the symptoms mentioned above, complications such as a severe pneumonia, acute respiratory distress syndrome (ARDS) kidney failure and fatal heart damage may develop. Dyspnea is one of the most prominent symptoms for COVID-19. Since COVID-19 affects the respiratory system, pulmonary rehabilitation has an important place in the treatment of patients. Dyspnea is one of the most prominent symptoms for COVID-19. Our clinical observations are of the opinion that dyspnea is observed even in patients with mild COVID-19 pneumonia. Applying deep breathing exercise with triflo in COVID-19 patients, can contribute to relieving dyspnea, reducing / eliminating anxiety, and increasing quality of life. In the light of this information, the aim of this study is to determine the effect of deep breathing exercise with triflo on dyspnea, anxiety and quality of life in patients with dyspnea who are hospitalized for COVID-19.

Research Hypotheses H1: Patients with COVID-19 pneumonia who undergo deep breathing exercise with triflo will have a lower dyspnea level than the patient group in which this exercise is not applied.

H2: Patients with COVID-19 pneumonia who underwent deep breathing exercise with triflo will have a lower anxiety level than the patient group in whom this exercise was not applied.

H3: Patients with COVID-19 pneumonia who underwent deep breathing exercise with triflo will have a higher quality of life than the patient group in whom this exercise was not applied.

DETAILED DESCRIPTION:
The world is facing an extremely important global epidemic. Coronavirus disease 2019 (COVID-19) epidemic, which first appeared in Wuhan, China in late 2019 and rapidly affected all countries of the world, was declared as a pandemic by the World Health Organization (WHO) on March 11, 2020. Coronavirus disease 2019 affects both the upper (i.e. sinuses, nose and throat) and lower (i.e. trachea and lungs) airways, causes respiratory tract diseases ranging from asymptomatic or cold to more severe lung diseases (Acute Respiratory Distress Syndrome-ARDS). COVID-19 has many symptoms. Dyspnea is one of the most prominent symptoms for COVID-19. The relationship between dyspneaand COVID-19 is not fully explained. Our clinical observations are of the opinion that dyspnea is observed even in patients with mild COVID-19 pneumonia.

Since COVID-19 affects the respiratory system, pulmonary rehabilitation has an important place in the treatment of patients. Deep breathing exercise applied within the scope of pulmonary rehabilitation expands the airways, facilitates gas exchange, increases the amount of oxygen reaching the cells, provides the release of tracheabronchial secretions, regulates the pulmonary circulation and thus increases the lung capacity. Deep breathing exercise also plays a role in lowering blood pressure and in reducing / relieving anxiety. Studies have stated that patients who are trained about deep breathing have better exercise status, that deep breathing exercise have increased systolic and diastolic blood pressure of and anxiety at statistically significant level. Triflo is a device that helps the patient to breathe deeply. It is seen as more advantageous in terms of use, as it provides visual information about the depth of breathing. The use of Triflo is used to support the determination of the patient's inspiration capacity, normal inspiration and deep breathing.

COVID-19, it has been determined that it improves respiratory function, quality of life and anxiety of the elderly and has little effect on depression.

The effects of COVID-19 disease on the lung and respiratory system appear to be quite serious. Since there is not enough information about the long-term results yet, its effect on patients and lungs after active period is not clearly known. The one of the most important data the investigators have now is that most of the patients experience dyspnea. In the literature, there has been no study examining the effect of respiratory exercise on dyspnea, anxiety and quality of life in patients diagnosed with COVID-19 pneumonia. However, applying deep breathing exercise with triflo in COVID-19 patients, can contribute to relieving dyspnea, reducing / eliminating anxiety, reducing / eliminating respiratory system complications, preserving / improving respiratory function, maintaining or increasing lung volume, accelerating recovery and increasing quality of life. In the light of this information, the aim of this study is to determine the effect of deep breathing exercise with triflo on dyspnea, anxiety and quality of life in patients with dyspnea who are hospitalized for COVID-19.

MATERIALS AND METHODS This single-centered, randomized controlled study will be held in Ankara city hospital in Turkey. Ethics committee approval was obtained from Ankara City Hospital Ethics Committee (Date:12/23/2020 Number:E.Kurul-E1-20-1403). The investigators also have received permission from the Ministry of Health of the Republic of Turkey for the study (Date:12/04/2020- Name and number: Hatice ÖNER CENGİZ-2020-12-04T12_09_16). Before the study, "enlightened informed consent" will be obtained from all participants. The entire study will be conducted in accordance with the Consolidated Standards of Reporting Trials (CONSORT) 2010 guidelines and directives.

Data will be collected between January 2021 and March 2021 from 44 patients treated at Ankara City Hospital COVID-19 clinics.

Randomized block assignment was used to assign 44 patients to the intervention group (n = 22) and the control group (n = 22). The investigators did block randomization, via a computer program (sealed envelope, https://www.sealedenvelope.com/ , randomization code: 34780089372265). A randomized block procedure (Vickers, 2006) was performed as follows: (a) a block size of 4 was selected; (b) subjects were calculated as having eleven conditions (ABBA, ABBA, BAAB, AABB, BAAB, BABA, AABB, BABA, ABBA, BABA and BAAB); and (c) blocks were randomly selected to determine the assignment of all 44 participants, with an allocation ratio of 1:1.

The investigators used the G*Power (Version 3.1.9) test to determine the sample size. In the analysis performed as a priori, The design of the study required a minimum sample size of 44 participants.

The data of the patient will be collected by the researchers by using the Patient Sociodemographic and Medical Data Form, Dyspnea-12 Scale, Beck Anxiety Inventory and SF-36 Short Form face-to-face and via telephone interviews. During the application of the scales, all measures will be taken to prevent virus spread.

Sociodemographic and Medical Data Form Sociodemographic and Medical Data Form prepared by the researchers consists of 14 questions including age, gender, marital status, education level, body mass index, presence of chronic disease, symptoms due to COVID-19 infection, experiencing dyspnea, frequency of dyspnea, factors affecting dyspnea, the number of respirations, oxygen saturation, blood gas analysis results.

Observation indicators:

Primary outcome: Oxygen saturation, respiratory assessment and dyspnea level Secondary outcomes: Anxiety and quality of life level

1. Oxygen saturation and respiratory rate: The respiratory rate of the patient and oxygen saturation from the fingertips of the patients will be evaluated by the researchers using the same pulse oximeter device.
2. Dyspnea: The dyspnea level of the patients will be evaluated with the Dyspnea-12 form. Dyspnea-12 scale consists of 2 sub-dimensions and a total of 12 items. The Turkish validity and reliability study of the scale was conducted in 2018, and its Cronbach's alpha reliability coefficient was found to be 0.97. Permission to use the scale has been obtained.
3. Anxiety: The anxiety level of the patients will be evaluated with the Beck Anxiety Inventory. Beck Anxiety Inventory is a scale developed in 1988 and used to determine the frequency of anxiety symptoms experienced by individuals. The Turkish validity and reliability study of the scale is available in the book "Clinical Scales Used in Psychiatry" and is widely used in studies conducted in our country.
4. Life quality: Life quality levels of patients will be evaluated with the World Health Organization Quality of Life Scale Short Form. The World Health Organization Quality of Life Scale Short Form is the abbreviation of World Health Organization Quality of Life Assessment (WHOQOL) scale, which was prepared to evaluate how the individual perceives the quality of life, consisting of 100-questions and reduced to 26 questions. The scale, which includes closed-ended questions, consists of four sub-domains: physical, social, environmental and psychological. The scale does not have a full score, and an increase in score indicates an improvement in quality of life. The Turkish validity and reliability study of the scale was conducted in 1999 and the number of questions was increased to 27 by adding a national question to the scale during their study.

Implementation of the initiative The investigators will include 22 patients in the intervention group, 22 patients in the control group and with the block randomization method, starting from the date the study was planned in this study. The investigators will obtain informed consent from patients who agreed to participate in the study and who meet the inclusion criteria. The investigators will monitor each patient until they are discharged. The investigators will exclude patients who were transferred to the intensive care unit or died during follow-up. All patients included in the study will receive all medical treatment administered in the hospital.

Interventions group. The investigators will apply a sociodemographic and medical data form, Dyspnea-12 scale, Beck Anxiety Inventory and SF-36 Short Form to 22 patients included in the intervention group on the first day of hospitalization. The investigators will give the triflo device to patients in the intervention group. The investigators will send the training video The investigators have prepared on how to apply the triflo deep breathing exercise to the patient's mobile phone to prevent virus spread and The investigators will ask the patient to do deep breathing with the triflo 5-10 times an hour by watching this video. The investigators will make the patients do the exercise through video calls, provide information on whether they are doing it right or not, and answer their questions. After the patients have breakfast in the morning, they will start their exercises and The investigators will make them do it 5-10 times an hour until they go to sleep. Until the patients are discharged, The investigators will evaluate respiratory rate, oxygen saturation with a pulse oximeter device without oxygen support and make them fill the Dyspnea-12 scale. The investigators will fill the Dyspnea-12 scale, Beck Anxiety Inventory and SF-36 Short Form while the patients are discharged.

Control group. The control group will comprise 22 patients treated for COVID-19 pneumonia at the hospital where the study was conducted. The investigatorswill make these patients fill the Sociodemographic and medical data form, Dyspnea-12 scale, Beck Anxiety Inventory and SF-36 Short Form at the beginning of the study; Dyspnea-12 scale every day until discharge ; the Dyspnea-12 scale, Beck Anxiety Inventory, and SF-36 Short Form during discharge.

Data will be evaluated with Statistical Package for Social Sciences 25 (SPSS) program using tests suitable for the distribution of data.

ELIGIBILITY:
Inclusion Criteria:

The patients,

* who are in clinical treatment for COVID-19 pneumonia;
* who are 18 years of age or older, mentally healthy;
* who can speak and understand Turkish;
* who owns and can use smartphones;
* who suffer from dyspnea,
* who do not have chronic diseases related to the respiratory system (lung diseases, heart diseases, etc.);
* who are volunteers, will be included in the study.

Exclusion Criteria:

The Patients

* for whom the data required for the study could not be collected;
* who are unable to complete the work (not wanting to continue working, transferred to the intensive care unit and died);
* who do not agree to participate in the study, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation (%) | until the treatment is completed,an average of 7 days
  Oxygen saturation (%) The oxygen saturation of the patient from the fingertips of the patients will be evaluated by the researchers using the same pulse oximeter device everyday.
Respiratory rate per minute | until the treatment is completed,an average of 7 days
  The respiratory rate of the patient will be evaluated by the researchers every day by counting the respiratory rate per minute.
Dyspnea level | until the treatment is completed,an average of 7 days
  The dyspnea level of the patients will be evaluated with the Dyspnea-12 form.Dyspnea-12 scale is a scale that measures the severity of dyspnea (shortness of breath) and consists of 2 sub-dimensions and a total of 12 items.

SECONDARY OUTCOMES:
Anxiety | post-treatment change (one week change)
  The anxiety level of the patients will be evaluated with the Beck Anxiety Inventory. Beck Anxiety Inventory is a scale developed by Beck et al. In 1988 and used to determine the frequency of anxiety symptoms experienced by individuals.The inventory is a Likert-type scale with 21 items scored between 0 and 3. The highest score that can be obtained from the scale is 63. A high total score indicates a high level of anxiety.
Quality of life level | post-treatment change (one week change)
  Life quality levels of patients will be evaluated with the World Health Organization Quality of Life Scale Short Form. The World Health Organization Quality of Life Scale Short Form is the abbreviation of World Health Organization Quality of Life Assessment (WHOQOL) scale, which was prepared to evaluate how the individual perceives the quality of life, consisting of 100-questions and reduced to 26 questions. The scale, which includes closed-ended questions, consists of four sub-domains: physical, social, environmental and psychological.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice ÖNER CENGİZ, Study Director — Ankara University
Locations (1):
- Hatice ÖNER CENGİZ, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigors do not intend to share research data with other researchers. The investigors may only share data from participants for meta-analysis study of randomized controlled trials.

REFERENCES:
- [Derived] Oner Cengiz H, Ayhan M, Guner R. Effect of deep breathing exercise with Triflo on dyspnoea, anxiety and quality of life in patients receiving covid-19 treatment: A randomized controlled trial. J Clin Nurs. 2022 Dec;31(23-24):3439-3453. doi: 10.1111/jocn.16171. Epub 2021 Dec 12. PMID 34897869